CLINICAL TRIAL: NCT06665685
Title: Using Gait Data to Inform Prescription Practice Among Nursing Home Residents to Reduce Medication-Induced Gait Disturbances
Brief Title: BioButton Among Nursing Home Residents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Charles Lin (Other)
Collaborators: Jewish Healthcare Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Charles Lin, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24050088
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Gait; Medication Induced Gait Disturbances

STUDY DESIGN:
Intervention Model Description: Study design will enroll arm 1 of 60 patients who will wear the device, BioButton, during their nursing home care. Arm 2 will consist of 10 nurses who have been assigned to care for one or more of the patients in Arm 1 to discuss device feasibility in terms of clinical care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Patient Group (Experimental): Patients in this arm will wear the device, BioButton, continuous for 30 days as it collects physiologic and gait data, while receiving otherwise routine, standard of care.
  Interventions: Device: BioButton Device
- Nurse Group (Experimental): Nurses caring for patients wearing the device, BioButton, will assist in placing and removing the device. Otherwise, they will provide routine, standard of care to the enrolled patients to determine the overall feasibility of the device for clinical care providers.
  Interventions: Device: Providing Clinical Care with BioButton Device

INTERVENTIONS:
Device: BioButton Device — BioButton is a remote wearable multi-parameter monitor, to identify gait disturbances that occur as a side effect of polypharmacy. This arm will be the patient wearing the device during their Nursing Home stay for 30-days.
  Arms: Patient Group
Device: Providing Clinical Care with BioButton Device — BioButton is a remote wearable multi-parameter monitor, to identify gait disturbances that occur as a side effect of polypharmacy. This arm will provide care for patients wearing the BioButton device during their Nursing Home stay for 30-days.
  Arms: Nurse Group

SUMMARY:
This pilot study will explore the use of the BioIntellisense BioButton, a remote wearable multi-parameter monitor, to identify gait disturbances that occur as a side effect of polypharmacy.

DETAILED DESCRIPTION:
By 2030, an anticipated seven adults over 65 years old are projected to die every hour from a fall in the United States. This highlights the growing percentage of the elderly in our population and the impact of falls on them. Nationally, over 25% of older adults report falling each year and falls are the leading cause of fatal and non-fatal injuries. In Pennsylvania, 30% of older adults report falling each year, an underreported value that can be as high as 60%. The cost of care for falls is over $50 billion annually in the United States according to the Centers for Disease Control (CDC). Nursing home residents are especially at risk; among nursing home residents, the risk of falling is 2x greater than community residents.

Nursing home residents who take multiple medications especially antidepressants, anxiolytics, and blood pressure drugs have an increased risk for falling. Polypharmacy especially the use of five or more medications is significantly associated with a 21% increase of falls. Unfortunately, gait data is not routinely collected or available to geriatric clinicians for making medication decisions. Empowering clinicians with gait data can be a powerful piece of the puzzle; this information may help them decide whether the benefit of starting a new anti-hypertensive or mood medication is worth the risk.

Clinicians informed with gait data can make better medication decisions for their elderly patients; they will be able to consider gait disturbance and fall risk in their clinical judgement. As a result, gait data from continuous wearable technology can adjust medication practices, and reduce medication-induced falls. Moreover, the concept for gait-informed prescription practice complements the 4Ms (what matters, medication, mentation, and mobility) employed by age-friendly health systems. Continuous gait data can inform the implementation of the 4Ms by (1) engaging patients and their families about their care priorities related medications and their impact on gait, (2) adjusting medications that affect mobility, and (3) addressing depression treatment with behavioral modifications instead of medications. Results from this project can inform future studies that will move the needle towards implementing care practices consistent with the 4Ms.

ELIGIBILITY:
Inclusion Criteria:

* Age >18yrs
* Presence of gait documentation in EMR

Exclusion Criteria:

* Age <18yrs
* Non-English-speaking patients
* Patients who cannot provide consent due to cognitive status
* Bedbound, unable to stand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Participant safety | 30-days
  This outcome measure will be reported via the % of patients who reported experiencing adverse events related to wearing the device (skin irritations, significant discomfort, etc.)
Protocol compliance | 30-days
  This outcome measure will be reported via the % of patients who were able to wear the device for the full 30-days.
Acceptability | 30-days
  This outcome measure will be reported via % of nurses who report that 'Yes' to the question: Would you recommend the patch to other nurses? on their acceptability survey.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Lin, MD, Principal Investigator — UPMC, University of Pittsburgh
Locations (1):
- UPMC Canterbury Place, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No